CLINICAL TRIAL: NCT00418028
Title: Randomized Phase II Trial of Continuous Versus Standard Capecitabine in Advanced Breast Cancer.
Brief Title: Standard Versus Continuous Capecitabine in Advanced Breast Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, Miguel Martin, MD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/237; 2004-002759-15 (EudraCT Number)
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Breast Cancer
Keywords: capecitabine; schedule; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Cint (Active Comparator): Capecitabine will be administered orally at a dose of 1250 mg/m2 twice-daily (in the morning and in the evening, the equivalent of a total daily dose of 2500 mg/m2) for 14 days, in 3 week cycles with a resting period of 7 days,until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
  Interventions: Drug: Capecitabine
- B Ccont (Experimental): Capecitabine 800 mg/m2 orally twice-daily (in the morning and in the evening the equivalent of one dose of 1600 mg/m2) for 21 days, in 3 week cycles without resting period, until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine
  Other Names: xeloda

SUMMARY:
Capecitabine is active in metastatic breast cancer but the conventional schedule (1250 mg/m2/12 hr 2 weeks on, one week off) produces grade 2 or greater hand and foot syndrome in up to 50% of patients leading to those reductions. There are theoretical reasons to administer S-phase specific agents in continuous, protracted rather than intermittent schedules. The investigators study compares the standard schedule (1250 mg/m2/12 hr 2 weeks on, one week off) with a continuous administration schedule (800 mg/m2/12hr). The latter administer approximately the same cumulative dose of capecitabine as the standard schedule. The study hypothesis is that grade 2 or greater hand and foot syndrome will be reduced from 50% (standard arm) to 20% (experimental arm). The investigators assume similar antitumor activity in both arms.

DETAILED DESCRIPTION:
Capecitabine is active in metastatic breast cancer but the conventional schedule (1250 mg/m2/12 hr 2 weeks on, one week off) produces grade 2 or greater hand and foot syndrome in up to 50% of patients leading to those reductions. Some authors have tested continuous administration schedules of capecitabine, showing better tolerance and apparently similar antitumor activity. Capecitabine is a pro-drug of 5-FU and mimics an i.v. continuous infusion administration of this antimetabolite. On the other hand, there are theoretical reasons to administer S-phase specific agents in continuous, protracted rather than intermittent schedules. Our study compares the standard schedule(1250 mg/m2/12 hr 2 weeks on, one week off)with a continuous administration schule (800 mg/m2/12hr). The latter schedule administer approximately the same cumulative dose of capecitabine as the standard one. The study hypothesis is that grade 2 or greater hand and foot syndrome will be reduced from 50% (standard arm) to 20% (experimental arm). The investigators assume similar antitumor activity in both arms.

ELIGIBILITY:
Inclusion Criteria

1. Patients diagnosed with metastatic breast cancer
2. Patients that either have received previous treatment with anthracyclines and/or taxanes or not (either as advance or in metastatic disease).
3. The patient is ambulatory with a functional ECOG < 2 status (see Appendix 2).
4. Patient presents, at least one lesion measurable according to RECIST criteria (see Appendix 3)
5. Patients with a life expectancy of at least 3 months.
6. Patients that agree to and are able to fulfill the requirements of the whole protocol through the whole study.

Exclusion criteria:

1. Patients that have previously shown unexpected severe reactions to therapy with fluoropyrimidines or with a known sensitivity to 5-fluorouracile.
2. Patients previously treated with capecitabine.
3. Patients with organ transplants.
4. Other diseases or severe affections:

   1. Patients with previous convulsions, central nervous system diseases or psychiatric diseases, including dementia, that the investigator might consider clinically significant and which adversely affect therapeutic compliance.
   2. Patients with severe intellectual impairment, unable to carry out basic daily routines and established depression.
   3. Clinical significant cardiac disease (e. g. . congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia not fully controlled with medication) or myocardial infarction within the last 12 months.
   4. Severe renal impairment (baseline creatinine clearance < 30 ml/min)
5. Patients with signs of metastasis in the CNS. Patients with a history of uncontrolled convulsions, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake should be excluded.
6. Patients with an active infection.
7. Patients with a history of other neoplasias during the previous five years, except for basal cell skin cancer or cervical cancer in situ, both cured.
8. Patients showing the following laboratory values:

   1. Neutrophil count < 555 x 109/l
   2. Platelet count< 100 x 109/l
   3. Serum creatinine > 1,5 x upper normality limit
   4. seric bilirubin > 2,0 x upper normality limit
   5. ALAT, ASAT > 2,5 x upper normality limit or > 5 x upper normality limit in case of liver metastases
   6. Alkaline phosphatase > 2,5 x upper normality limit > 5 x upper normality limit in case of liver metastases o > 10 x upper normality limit in case of bone metastases.
9. Patients under radiotherapy four weeks prior to the initiation of the study treatment, or under previous radiotherapy on the marker lesions be measured during the study (new marker lesions that appear in previously irradiated areas are accepted) or patients who are receiving programmed radiotherapy.
10. Patients under major surgery within 4 weeks prior to study treatment or who have not completely recovered from the effects of major surgery.
11. Patients who lack upper gastrointestinal tract physical integrity or with malabsorption syndrome.
12. Patients who have received more than two cycles of chemotherapy for the metastatic disease.
13. Patients Her2 + per FISH ó +++ Immunohistochemistry

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2005-09; Primary Completion 2011-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Martin, MD,PhD, Study Chair — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

REFERENCES:
- [Derived] Martin M, Martinez N, Ramos M, Calvo L, Lluch A, Zamora P, Munoz M, Carrasco E, Caballero R, Garcia-Saenz JA, Guerra E, Caronia D, Casado A, Ruiz-Borrego M, Hernando B, Chacon JI, De la Torre-Montero JC, Jimeno MA, Heras L, Alonso R, De la Haba J, Pita G, Constenla M, Gonzalez-Neira A. Standard versus continuous administration of capecitabine in metastatic breast cancer (GEICAM/2009-05): a randomized, noninferiority phase II trial with a pharmacogenetic analysis. Oncologist. 2015 Feb;20(2):111-2. doi: 10.1634/theoncologist.2014-0379. Epub 2015 Jan 19. PMID 25601966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2004 and August 2010, 195 patients were randomly assigned to Cint (97) and Ccont (98) in 13 GEICAM sites in Spain.
Groups:
- Arm A (Cint): Capecitabine will be administered orally at a dose of 1250 mg/m2 twice-daily (in the morning and in the evening, the equivalent of a total daily dose of 2500 mg/m2) for 14 days, in 3 week cycles with a resting period of 7 days,until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
  capecitabine: 1250 mg/m2 twice a day orally x 14 days every 3 weeks until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
- Arm B (Ccont): Capecitabine 800 mg/m2 orally twice-daily (in the morning and in the evening the equivalent of one dose of 1600 mg/m2) for 21 days, in 3 week cycles without resting period, until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
  drug: capecitabine: 800 mg/m2 twice a day orally continuous administration until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
Period: Overall Study
Arm/Group | Arm A (Cint) | Arm B (Ccont)
Started | 97 | 98
Completed | 95 | 97
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Cint) | Arm B (Ccont) | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 65 | 120
  >=65 years | 42 | 33 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.07 (13.21) | 58.59 (11.66) | 59.82 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 98 | 195
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 97 | 98 | 195

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to Progression (TTP) is defined as the time (in months) from the moment the patient starts the study treatment to the date of progressive disease. That is, a patient has an event is she progresses or dies due to progressive disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0).
Time Frame: After 1 year from the treatment start day.
Population: A total of 192 patients (95 in Arm A and 97 in Arm B) were considered for this analysis but 36 were censored (23 in Arm A and 13 in Arm B). Patients censored are those that did not progress or die due to progressive disease during the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A (Cint): Capecitabine will be administered orally at a dose of 1250 mg/m2 twice-daily (in the morning and in the evening, the equivalent of a total daily dose of 2500 mg/m2) for 14 days, in 3 week cycles with a resting period of 7 days,until disease progression or severe toxicity.
- Arm B (Ccont): Capecitabine 800 mg/m2 orally twice-daily (in the morning and in the evening the equivalent of one dose of 1600 mg/m2) for 21 days, in 3 week cycles without resting period, until disease progression or severe toxicity.
Arm/Group | Arm A (Cint) | Arm B (Ccont)
Number analyzed (Participants) | 72 | 84
months | 8.68 [6.55 to 11.05] | 6.84 [6.02 to 8.06]
Statistical Analysis 1: Comparison: Arm A (Cint) vs Arm B (Ccont); Test type: Non-Inferiority or Equivalence — If we assume that the non-inferiority level is up to 15% lower (equivalent to a median progression-free time of 3 months), for a one-sided error α=0.05, and 80% power, are necessary 88 patients per group. Considering an dropout rate of around 10%, the number of patients would be 98 per group; p = 0.1224, Log Rank; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.9 to 1.7]

2. Secondary Outcome: Response Rate
Description: Response was evaluated using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), every 3 cycles of chemotherapy (each cycle lasts 3 weeks) and at the end of treatment (at 21 weeks from the start of treatment).
Time Frame: Through the study treatment, an average of 5 months.
Population: There were 95 patients in Arm A and 97 patients in Arm B. There were 13 patients without response evaluation (9 in Arm A and 4 in Arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cint) | Arm B (Ccont)
Number analyzed (Participants) | 86 | 93
Participants | 30 | 31
Statistical Analysis 1: Comparison: Arm A (Cint) vs Arm B (Ccont); Test type: Superiority; p = 0.8269, Chi-squared

3. Secondary Outcome: Response Duration
Description: Response duration is computed for all patients with Partial Response or Complete Response, during the treatment period, as the time from the moment the Partial or Complete Response is reported to the date the patient Progresses or Dies, whichever happens first.
  A patient is censored if she does not progress or die. In these cases Response duration is computed as the time from the moment the Partial or Complete Response is reported to the last contact date.
Time Frame: Time from the moment the Partial or Complete Response is reported to the date the patient Progresses or Dies, whichever happens first, assessed up to 72 weeks.
Population: From 192 patients (95 in Arm A and 97 in Arm B), 61 patients had Complete Response or Partial Response (30 in Arm A and 31 in Arm B).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Cint) | Arm B (Ccont)
Number analyzed (Participants) | 30 | 31
Months | 10.07 [7.96 to 16.71] | 7.20 [4.11 to 12.7]
Statistical Analysis 1: Comparison: Arm A (Cint) vs Arm B (Ccont); Test type: Superiority; p = 0.5703, Log Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.67 to 2.07]

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (TTF) is defined as the time (in months) from the moment the patient starts the study treatment to the end of treatment date (due to death, progressive disease, adverse events, patient's decision or investigator criteria.
  If a patient did not end the treatment, it is censored. The censoring date is the date of the last dose received.
Time Frame: Time (in months) from the moment the patient starts the study treatment to the end of treatment date (due to death, progressive disease, adverse events, patient's decision or investigator criteria, assessed up to 72 months.
Population: This outcome only was analyzed in the Per Protocol Population (182 patients).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Cint) | Arm B (Ccont)
Number analyzed (Participants) | 90 | 92
Months | 5.41 [4.34 to 8.03] | 5.87 [3.55 to 7.14]
Statistical Analysis 1: Comparison: Arm A (Cint) vs Arm B (Ccont); Test type: Superiority; p = 0.4676, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.83 to 1.50]

5. Secondary Outcome: Overall Survival
Description: An event is defined as death. A patient is censored if she does not die. The censoring date is last contact date.
Time Frame: Time to survival is the number of months from the study treatment start date to the date of death, assessed up to 100 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Cint) | Arm B (Ccont)
Number analyzed (Participants) | 95 | 97
Months | 27.34 [22.40 to 32.11] | 24.11 [18.16 to 33.06]
Statistical Analysis 1: Comparison: Arm A (Cint) vs Arm B (Ccont); Test type: Superiority; p = 0.5688, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.66 to 1.25]

6. Secondary Outcome: Clinical Benefit
Description: A patient experiences a Clinical Benefit if the following is satisfied:
  Criterion: The patient has "Complete response", "Partial Response" or "Stable Disease" and it continues during more than 3 months.
Time Frame: Months from "CR","PR" or "SD" (the first one) until Progression date, new treatment or last contact date.
Population: Only 179 patients had tumor evaluation data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Cint) | Arm B (Ccont)
Number analyzed (Participants) | 86 | 93
Participants | 56 | 56
Statistical Analysis 1: Comparison: Arm A (Cint) vs Arm B (Ccont); Test type: Superiority; p = 0.4984, Chi-squared

7. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as the time (in months) from the moment the patient starts the study treatment to the date of progressive disease. That is, a patient has an event is she progresses or dies for any reason.
Time Frame: Time (in months) from the moment the patient starts the study treatment to the date of progressive disease assessed up to 84 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Cint) | Arm B (Ccont)
Number analyzed (Participants) | 95 | 97
Months | 8.52 [5.66 to 10.20] | 6.84 [6.02 to 8.06]
Statistical Analysis 1: Comparison: Arm A (Cint) vs Arm B (Ccont); Test type: Superiority; p = 0.2556, Log Rank; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.88 to 1.63]

ADVERSE EVENTS:
Time Frame: During the study treatment (Metastatic Breast Cancer patients), up to 30 weeks approximately.
Groups:
- A Cint: Capecitabine will be administered orally at a dose of 1250 mg/m2 twice-daily (in the morning and in the evening, the equivalent of a total daily dose of 2500 mg/m2) for 14 days, in 3 week cycles with a resting period of 7 days,until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
  drug: capecitabine: 800 mg/m2 twice a day orally continuous administration until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
- B Ccont: Capecitabine 800 mg/m2 orally twice-daily (in the morning and in the evening the equivalent of one dose of 1600 mg/m2) for 21 days, in 3 week cycles without resting period, until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
  capecitabine: 1250 mg/m2 twice a day orally x 14 days every 3 weeks until disease progression or severe toxicity. Dose adjustments were made in patients with grade 3 or greater diarrhea or hand and food syndrome.
Arm/Group | A Cint | B Ccont
Serious Adverse Events (participants affected / at risk) | 13/95 | 4/97
Other Adverse Events (participants affected / at risk) | 81/95 | 51/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A Cint (N=95) | B Ccont (N=97)
Diarrhea (Gastrointestinal disorders) | 6 | 0
Febrile neutropenia (Infections and infestations) | 2 | 0
Obstruction (Gastrointestinal disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Mucositis/stomatitis (Gastrointestinal disorders) | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 | 1
Infection with unknown ANC (Infections and infestations) | 0 | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A Cint (N=95) | B Ccont (N=97)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 39 | 41
Grade 3-4 Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Grade 3-4 Neutropenia (Blood and lymphatic system disorders) | 9 | 2
Grade 3-4 Diarrhea (Gastrointestinal disorders) | 19 | 6
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 11 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days